CLINICAL TRIAL: NCT06955728
Title: A Phase-IV Individually Randomized, Placebo-controlled Trial on Safety of RSVA/B-preF Vaccine in Pregnant Women and Efficacy Against Severe RSV-associated Lower Respiratory Tract Infection in Infants
Brief Title: A Clinical Trial on Safety in Pregnant Women and How Well the Infant is Protected Against RSV-associated Lower Respiratory Tract Infection When the Pregnant Woman Receives the Approved RSV Vaccine Compared to a Placebo.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: World Health Organization (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RSV_IMPACT
Record Dates: First submitted 2025-04-14; First posted 2025-05-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: RSV Infections; RSV Immunisation; Preterm Labour
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Obstetric Labor, Premature | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Control group will receive the placebo which will match the vaccine to maintain the blind but will not contain any active product. Participants will be randomised 1:1
  Interventions: Other: Placebo
- ABRYSVO (RSV A/B-pre-F vaccine) (Active Comparator): ABRYSVO vaccine developed by Pfizer. The active ingredients in RSVpre-F are 2 stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B, in a lyophilized dosage form for reconstitution
  Interventions: Drug: Vaccine

INTERVENTIONS:
Drug: Vaccine — The active ingredients in RSVpreF are 2 stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B, in a lyophilized dosage form for reconstitution.
  Arms: ABRYSVO (RSV A/B-pre-F vaccine)
Other: Placebo — Placebo matched to vaccine but not containing any active ingredients
  Arms: Placebo

SUMMARY:
Respiratory syncytial virus (RSV) is a virus that often affects children during childhood. Even though most cases of RSV are mild, it can cause serious disease and even death - especially in very young babies, babies born too early and those born with heart and lung problems. It is the most common cause for children under 5 years old to be hospitalised. In 2019, there were about 33 million RSV-infections in the lower respiratory tract (in the lungs and below the voice box) of which 3,6 million people were hospitalised and 26,300 passed away in hospital due to RSV. Almost half (50%) of deaths that are caused by RSV, happen in children younger than 6 months old and the majority (more than 95%) of these deaths happen to infants and children in low- and middle-income countries.

A way that can help protect babies from becoming infected is through giving vaccines against the germ (RSV) that is targeted for prevention. There are currently no registered vaccines that can be given directly to babies however there is a lot of information available that shows that a vaccine can be safely giving to a mother while she is still pregnant. The mother then produces antibodies (protection cells) that is transferred to the baby before the baby is born, and the baby is protected from getting sick during the first few months of life.

One of the vaccines that has been developed (ABRYSVO) has been used in many clinical trials in pregnant moms (and older people) to test if it is safe and will protect young babies and much older people who are all at the highest risk for a severe RSV disease. The vaccine was given to more than 4,000 pregnant women. The results from the study and previous studies showed that the vaccine was safe and the babies had a lower chance of getting severe RSV disease and going to hospital. It showed that the vaccine prevented severe RSV infection in around 80% of babies younger than 90 days, and 70% of babies younger than 6 months. Therefore, the vaccine has been licensed in a few countries around the world (including the United States of America and other high-income countries) which means that pregnant women can receive this vaccine during their pregnancy if they wish to (without being on a clinical trial). It has also been licensed in South Africa but is not yet available in the country for pregnant women to receive. The licensure is also underway in other African countries.

However, the results of the previous studies of this vaccine also showed that a slightly higher number of premature babies were born to women who received the vaccine compared to women who did not receive the vaccine. The information received from these studies was however not enough to decide if the earlier births were related to the vaccine or not, and more information is needed - which is one of the main reasons for this study. Importantly, all of the babies who were born earlier were only born a few weeks earlier than expected (around 35 weeks of pregnancy), and all the babies were well and survived. The previous studies on this vaccine happened during the COVID-19 pandemic at which time people were wearing masks and contacting other people less therefore not spreading RSV around as we would normally expect. By doing this study, it will assist the investigators to determine if the vaccine is really as good as it is perceived to be for preventing serious RSV illness in the babies.

This RSV vaccine is a very important medical intervention, and it is as important that the effect that this vaccine will have on pregnant women and on the infants born to mothers who receive the vaccine can be measured. It is especially important in African and lower-middle income countries as the vaccine was not tested as much in people living in Africa compared to others. Therefore, the main reason for doing this trial is to see how much value the vaccine can bring to these countries in terms of protecting young babies and infants where many may get a severe infection and be hospitalised. It will also measure if the vaccine does increase the chances of a baby being born earlier than expected. It will only be carried out in the countries after the vaccine has been approved for use by pregnant women (at the right time) as part of their pregnancy care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women considered to be legally competent, as per country legislation, to consent for trial participation for herself and her newborn
* Gestational age ≥ 28wk0days to <36wks0days as per GAIA LOC criteria 1 to 2B who are not in active labour
* Mother is able to understand and comply with planned trial procedures
* Mother is attending ante-natal clinic
* Mother has documented test for HIV and syphilis during the current pregnancy,
* Provides written informed consent prior to initiation of trial. If the maternal participant is illiterate, a witnessed thumb-printed informed consent is acceptable
* Intention to deliver at a hospital or birthing facility where trial procedures can be obtained (for immunogenicity cohort)
* Expected to be available for the duration of the trial and can be contacted by telephone or by physical visit during trial participation
* Participant is willing to give informed consent for her infant to participate in the trial

Exclusion Criteria:

* Body mass index of >40 kg/m2 at the time of the first obstetric visit during the current pregnancy
* Bleeding diathesis or condition (past or present) associated with prolonged bleeding that would, in the opinion of the investigator, contra-indicate intramuscular injection
* History of severe adverse reaction associated with a vaccine
* Current pregnancy complications or abnormalities at the time of consent that will increase the risk associated with the participation in and completion of the trial, including but not limited to the following:

  1. More than two fetuses (i.e. twins will be allowed)
  2. Preeclampsia, eclampsia, or uncontrolled gestational hypertension
  3. Placental abnormality.
  4. Polyhydramnios or oligohydramnios
  5. Endocrine disorders, including untreated hyperthyroidism or untreated hypothyroidism, or uncontrolled diabetes mellitus at the time of consent.
  6. Any signs of premature labour with the current pregnancy or having ongoing intervention (medical/ surgical) in the current pregnancy to prevent preterm birth.
* At least THREE prior pregnancy complications or abnormalities at the time of consent, based on the investigator's judgment, that will increase the risk associated with the participation in and completion of the trial, including but not limited to the following:

  1. Prior preterm delivery between 18 to ≤34 weeks gestation, or birth weight <2200 grams.
  2. Prior stillbirth or neonatal death within 7 days of birth.
  3. Previous infant with a known genetic disorder or major congenital anomaly
* Mother who is positive for syphilis and untreated at time of enrolment
* Mother living with HIV/AIDS considered to have WHO Clinical Stage 3 or 4 AIDS, or considered to be clinically unstable
* Major illness of the maternal participant or conditions of the foetus that, in the investigator's judgment, will substantially increase the risk associated with the maternal participant's participation in, and completion of, the trial
* Congenital or acquired immunodeficiency disorder, or rheumatologic disorder or other illness requiring chronic treatment with known immunosuppressant medications, including monoclonal antibodies, within the year prior to enrolment
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behaviour or laboratory abnormality that may increase the risk associated with trial participation and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial
* Participation in other studies involving investigational drug(s) within 28 days prior to consent and/or during trial participation.
* Use of systemic corticosteroids for >14 days within 28 days prior to trial enrolment. Prednisone use of <20 mg/day for ≤14 days is permitted. Inhaled/nebulized, intra-articular, intra-bursal, or topical (skin or eyes) corticosteroids are permitted
* Current alcohol abuse or illicit drug use
* Receipt of blood or plasma products or immunoglobulin (Ig) in past 60 days or planned receipt through delivery, with exception of Rho(D) immune globulin (eg, RhoGAM), which can be given at any time
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during trial participation

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of RSVA/B-preF against RSV-A or RSV-B subtype confirmed severe LRTI through to 180 days of age by measuring the first occurrence of RT-PCR confirmed RSV severe LRTI | From infant birth to 180 days of age
  The presence of LRTI will be confirmed according to case definition. The severity of LRTI will be based on the WHO grading criteria
Evaluate the safety of RSVA/B-preF in relation to preterm births in women with gestational age (GA) staging Level of Certainty [LOC] 1 to 2B at time of enrolment by measuring the occurrence of preterm births (<37 weeks GA) | At delivery of the infant
  The GA staging will be based on Global Alignment on Immunization safety Assessment (GAIA) criteria

SECONDARY OUTCOMES:
Evaluate the efficacy of RSVA/B-preF against RSV-confirmed severe LRTI through to 90, 120 and 150 days of age by measuring the first occurrence of RT-PCR confirmed RSVA or RSVB severe LRTI | 90, 120 and 150 days of age
Evaluate the efficacy of RSVA/B-preF against RSV-confirmed LRTI resulting in hospitalization with use of supplemental oxygen OR O2 saturation of <92% (at 180 days, 90, 120 & 150 days) by measuring the first occurrence of RT-PCR confirmed RSVA or RSVB | At 90, 120, 150 and 180 days of age
Evaluate the efficacy of RSVA/B-preF against RSV-confirmed MA-LRTI and very-severe LRTI (at 180 days, and 90, 120 and 150 days) by measuring the first occurrence of RT-PCR confirmed RSVA or RSVB MALRTI or very-severe LRTI | 90, 120, 150 and 180 days of age
Evaluate the efficacy of RSVA/B-preF against RSV-confirmed: a. MA-LRTI; b. severe-LRTI; c. very-severe LRTI; d. LRTI hospitalization from 0 to 90 days and 91-180 days by measuring the first occurrence of RT-PCR confirmed RSVA or RSVB MA-LRTI | 0-90 and 91-180 days of age
Evaluate the efficacy of RSVA/B-preF against all-cause: a. MA-LRTI; b. severe LRTI; c. very-severe LRTI; d. LRTI hospitalization, by measuring the first occurrence of all-cause MALRTI | at 180 days, and 90, 120, and 150 days; and at 0-90 days and 91-180 days of age
Evaluate the safety of RSVA/B-preF against prematurity in women vaccinated at 28 to <32 weeks, 32 to 36 weeks by measuring the occurrence of pre-term delivery (<37 weeks) | At delivery of the infant
  Limited to women with GA staging using GAIA LOC 1 to 2B at time of enrolment
Evaluate the safety of RSVA/B-preF against prematurity occurring at 28 to <32 weeks, 32 to 36 weeks by measuring the occurrence of pre-term delivery in the mentioned intervals | At delivery of the infant
  Limited to women with GA staging using GAIA LOC 1 to 2B at time of enrolment
Evaluate the safety of RSVA/B-preF against low birth weight (<2500 grams) and very low birth weight (<1500 grams) by measuring the occurrence of low and very low birth weights | At delivery of the infant

CONTACTS AND LOCATIONS:
Overall Officials: Shabir Madhi, Study Chair — Wits Vaccines & Infectious Diseases Analytics Research Unit; Ziyaad Dangor, Study Director — Wits Vaccines & Infectious Diseases Analytics Research Unit
Locations (5):
- South Africa (5):
  - Wits RHI Shandukani CRS, Hillbrow, Gauteng
  - VIDA Nkanyezi Research Unit, Johannesburg, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - Wits Vaccines & Infectious Diseases Analytics (VIDA) Research unit, Soweto, Gauteng
  - MRC Unit on Child and Adolescent Health, Rondebosch, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Progress reports for this trial will be made available to the trial funder, ethics committees, regulatory authorities and other stakeholders. Final trial results will be shared with the same stakeholders within 3 months of final lock of the trial database. Study data will be shared with Pfizer in the event of safety concerns or a request from a regulatory agency. Manuscript(s) will be prepared and submitted for peer-review in open access journals. All proposed publications will first be reviewed by Pfizer prior to publication for review of potential confidential information. A publication plan and proposal for criteria of authorship will be established with the sites. The trial database will be made publicly available upon request. Any transfer of data, will be governed, by the terms of the local Ethics Committee (HREC).
Supporting Information: CSR, Analytic Code
Time Frame: Within 12 months of availability of study report
Access Criteria: Any transfer of data, will be governed, by the terms of the local Ethics Committee (HREC). Data sharing will be done on a collaborative basis, with the site PI (or his nominee) being included in any further interrogation of the data.